CLINICAL TRIAL: NCT05396820
Title: Adaptation of the Motor System to Experimental Pain
Acronym: KinesioPoint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universite du Littoral Cote d'Opale (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-A00271-42
Record Dates: First submitted 2022-05-18; First posted 2022-05-31 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Kinesiophobia; Pain, Acute
Keywords: kinesiophobia; experimental pain; corticospinal excitability; motor control; CUSOM
MeSH Terms: conditions — Kinesiophobia; Acute Pain

STUDY DESIGN:
Intervention Model Description: Cross sectional study
Masking Description: A randomized number is allocated for all participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental pain (Experimental): Experimental pain will be induced at the level of the dominant delto-pectoral groove of the participant (between the shoulder stump and the pectoral).
  Interventions: Other: Experimental pain

INTERVENTIONS:
Other: Experimental pain — Experimental pain will be induced by capsaicin 1% on intact, non-irritated and dry shoulder's skin. For the purposes of this study, we will remove this patch before the recommended application time in order to generate a pain. The participant will be seated on a chair facing a table so that his or her dominant forearm rests on the table. Markers will be placed at the table and chair legs as well as on the table, corresponding to the two support points of the elbow and the index finger, in order to standardize the starting position. The target of the pointing movement will be placed at 80% of this maximum distance. The investigator will tell the participant to stand by, and then, within 4 to 10 seconds, an audible signal will indicate to the subject that he/she should perform the pointing movement. The procedure will repeat after a 4-10 second pause. For each session, 30 pointing movements reaching the target will be performed.

SUMMARY:
This study aims to measure the impact of an experimental pain on electromyography, kinematics of motion and motor cortical excitability.

DETAILED DESCRIPTION:
The main objective of this study will be to determine if the influence of pain on the corticospinal excitability of M1 (via the slopes of the I/O curves) is dependent on the level of kinesiophobia.

The secondary objectives are firstly to measure the modifications induced by experimental pain on muscle activation synergies. Secondly, to measure the modifications induced by an experimental pain on the kinematics of the movement during a pointing task during the application of the pain. Finally, to determine if an experimental pain modifies the electrical activity of muscles located in the painful area during a pointing movement and the value of the cumulative sums (CUSUMs).

Inclusion Criteria:

* Males and females of legal age.
* Healthy subjects (who do not have self-reported neurological disorders)
* Subjects who have signed an informed consent (who have a good command of French)
* Subjects who are affiliated with or benefit from a social security plan

Criteria for non-inclusion:

* Psychiatric history obtained by physician questioning: individuals with mental retardation or severe impairment of cognitive, behavioral, or affective functions precluding understanding the protocol and signing informed consent
* Neurological history (epilepsy, stroke, surgeries performed on the brain or spinal cord, and history of neurological diseases affecting motor skills and sensation)
* Subjects who are unable to receive informed information (dementia, hearing problems, poor French proficiency, etc.)
* Contraindications to MST (epilepsy, intracranial metal foreign bodies, hearing aids or cochlear implants)
* Taking psychotropic medications
* Persons under guardianship or conservatorship
* Pregnant and nursing women
* Subjects with pacemakers

Assessment before pain induction:

► Corticospinal excitability of M1: The TMS will be used to establish the input-output (I/O) curves. Stimuli of variable intensity between the threshold value (or MT for motor threshold) and the maximum will be delivered. In total, about ten stimulation intensities will be tested, and for each stimulation intensity, ten stimuli will be delivered, allowing then to calculate the average of the MEPs in order to draw the I/O curves of each participant. As recalled by national and international recommendations, TMS is a noninvasive and painless technique whose use in the scientific literature is extremely abundant.

► Pointing task: The participant will be seated on a chair facing a table so that his or her dominant forearm rests on the table. Markers will be placed at the table and chair legs as well as on the table, corresponding to the two support points of the elbow and the index finger, in order to standardize the starting position. The index finger should be positioned on the midline. The maximum amplitude of the pointing movement on the median line will be determined and then the target of the pointing movement will be placed at 80% of this maximum distance. The investigators chose a single target so that reaction time would not be impacted by too much cognitive load. The investigator will tell the participant to stand by, and then, within 4 to 10 seconds, an audible signal ("beep") will indicate to the subject that he/she should perform the pointing movement. Then the subject will return to the starting position at rest, and the procedure will repeat after a 4-10 second pause. For each evaluation session, 30 pointing movements reaching the target will be performed, the first three of which will not be counted (familiarization). The kinematic parameters of the pointing movements will be recorded using a 3D motion analysis video system. The markers will be placed on C7, and on the dominant side on the acromion, the olecranon, the dorsal aspect of the wrist and on the distal phalanx of the index finger.

► Muscle activation synergies: To measure muscle activations during this pointing task, surface EMG recording of the anterior deltoid and upper trapezius muscles will be performed on the dominant upper limb using a wireless collection system. Raw data of kinematic and EMG parameters will be stored and processed offline. Trials where the reaction time is less than 100ms will be excluded from the analysis.

Assessment during experimental pain:

► Experimental Pain Induction: In this study, the application of a capsaicin 1% patch will be performed at the participant's dominant delto-pectoral groove (between the shoulder stump and pectoral) on intact, non-irritated, dry skin to generate experimental pain. For the purposes of this study, the investigators will remove this patch before the recommended application time (60 minutes) in order to generate a limited pain of 3 to 5/10 on a visual analog scale (VAS).

► Completion of the EKT-CF questionnaire: During the time of onset and stabilization of pain induced by the capsaicin 1% patch, the participant will be asked to complete the EKT-CF questionnaire in computerized form. An evaluation of the pain will be made at this time using a VAS and the value will be noted.

► TMS, Pointing and muscles activation: Once the pain has settled and stabilized, TMS, surface EMG and kinematic measurements will be performed again in the same way as described previously. The similar optimum stimulation point used for the TMS will be rigorously stimulated using the coordinates recorded previously.

The duration of the experimental session is estimated at 2h30min, distributed as follows: Information, eligibility and consent collection: 15 minutes; preparation of the experiment (installation of the electrodes, setting of the devices: 45 minutes; recordings: 90 minutes).

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects (who do not have self-reported neurological disorders)
* Subjects who have signed an informed consent (who have a good command of French)
* Subjects affiliated with or receiving social security benefits

Exclusion Criteria:

* Psychiatric history obtained through physician questioning: individuals with mental retardation or severe impairment of cognitive, behavioral, or emotional function that precludes understanding the protocol and signing informed consent
* Neurological history (epilepsy, stroke, surgeries performed on the brain or spinal cord, and history of neurological diseases affecting motor skills and sensation)
* Subjects who are unable to receive informed information (dementia, hearing problems, poor French proficiency, etc.)
* Contraindications to MST (epilepsy, intracranial metal foreign bodies, hearing aids or cochlear implants)
* Taking psychotropic medications
* Persons under guardianship or conservatorship
* Pregnant and nursing women
* Subjects with pacemakers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Corticospinal excitability | 1 hour
  It will be measured using transcranial magnetic stimulation at different intensities in order to model I/O curves for each participant. Measurements will be taken before (pain-free condition) and after (pain condition) the application of a patch of capsaicin 1%, at the shoulder. Electromyographic signals, induced by the magnetic stimuli, will be captured with surface electrodes glued to the skin the anterior deltoid and upper trapezius muscles. To facilitate obtaining deltoid MEPs, participants will be asked to voluntarily contract 8-12% of their maximum voluntary contraction. The Boltzmann sigmoidal function will be used to fit the data points to construct the I/O curves. The mathematical modeling of the I/O curves allows the calculation of three parameters: the slope, the plateau, and the S50, the intensity allowing to obtain a response twice less than the maximum response. These 3 parameters will be used to compare them with the 2 conditions (before and after pain).
Kinesiophobia | 5 minutes
  Kinesiophobia will be assessed using the French-Canadian version of the Tampa Kinesiophobia Questionnaire (EKT-CF). It takes the form of a self-reported questionnaire of 17 items using a Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree), with an acceptable degree of internal consistency (Cronbach's alpha = 0.71), satisfactory construct validity, and high sensitivity to change (intra-class correlation coefficient > 0.7). The total score is obtained by adding the value of the responses and is between 17 and 68. The value of 40/68 is considered as the threshold value at which kinesiophobia becomes significant.

SECONDARY OUTCOMES:
Activation synergies | 1 hour
  Surface electromyogram recordings of the anterior deltoid and upper trapezius muscles will be made on the dominant upper limb performing a pointing task and on which the experimental pain will be induced (pre-post measurements).
  The activation synergies will be recorded (relative durations between the onset of different surface EMG puffs of the targeted muscles).
Kinematic parameters: Linearity of motion | 1 hour
  Trajectory length ratio (TLR), defined as the ratio of the total length of the trajectory traveled by the hand divided by the shortest length between the start and end points. A ratio of 1 indicates an ideal trajectory; as the ratio increases, the trajectory becomes less direct.
Kinematic parameters: Smoothness of motion | 1 hour
  The number of velocity peaks on the kinematic path of the index. The higher this number, the less regular the motion.
Kinematic parameters: Maximum directional error | 1 hour
  Maximum orthogonal distance between the hand position and the straight line connecting the start and end points.
EMG data and cumulative summation: The area of the puffs | 1 hour
  The value of the area under the curves between the beginning and the end of the puffs.
EMG data and cumulative summation: CUSUMs | 1 hour
  The value of the CUSUMs of each puff, which represents the small variations that may appear in surface EMG and may be masked by background fluctuations.

CONTACTS AND LOCATIONS:
Locations (1):
- Eurasport, Loos, Nord, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duport A, Morel P, Leonard G, Devanne H. The influence of pain and kinesiophobia on motor control of the upper limb: how pointing task paradigms can point to new avenues of understanding. Pain. 2024 Sep 1;165(9):2044-2054. doi: 10.1097/j.pain.0000000000003213. Epub 2024 Mar 13. PMID 38501987